CLINICAL TRIAL: NCT06202339
Title: A Feasibility and Safety Study of Intratumoral Diffusing Alpha Radiation Emitters for the Treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva
Brief Title: Alpha Radiation Emitters Device for the Treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva (DaRT).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alpha Tau Medical LTD. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-VUL-01
Record Dates: First submitted 2023-12-31; First posted 2024-01-11 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2023-12

CONDITIONS: Carcinoma of the Vulva; Recurrent Carcinoma of the Vulva
Keywords: Cancer; Alpha emitting radiation; Brachytherapy; DaRT
MeSH Terms: conditions — Vulvar Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DaRT Seeds (Experimental): Intratumoral Diffusing alpha-emitters Radiation Therapy (DaRT) Seeds
  Interventions: Device: DaRT seeds

INTERVENTIONS:
Device: DaRT seeds — An intratumoral insertion of a seed(s), loaded with Radium-224, securely fixed in the seeds. The seeds release by recoil into the tumor short-lived alpha-emitting atoms

SUMMARY:
A unique approach for cancer treatment employing intratumoral diffusing alpha radiation emitter device for the treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva.

DETAILED DESCRIPTION:
This is an prospective Open label, single arm, multi center, interventional study treatment of Primary and Recurrent Squamous Cell Carcinoma of the Vulva .The study objectives are to collect data on the Feasibility and Safety of DaRT among patients who do not fit the entry of existing investigational trials.

The primary endpoint of the study is to evaluate the feasibility and safety of the Alpha DaRT sources for the treatment of vulva SCC. Feasibility will be determined according to the rate of successful placement of Alpha DaRT . Safety will be determined according to the overall incidence of device related AEs and SAE's graded according to CTCAE v5.0 criteria.

The Secondary endpoint of the study will be to evaluate efficacy, as determined by local control evaluation according to RECIST v1.1

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed newly diagnosed or recurrent (local) vulva SCC with or without distant metastases within 12 months
2. Tumor size ≤ 7 centimeters in the longest diameter.
3. Targeted lesion must be technically amenable for complete coverage (including margins) by the Alpha DaRT sources.
4. Measurable target according to RECIST v1.1
5. Interstitial implant indication validated by multidisciplinary team.
6. ECOG Performance Status ≤3.
7. Life expectancy ≥6 months.
8. Women Age ≥18
9. Willing and have the ability to provide signed Informed Consent.
10. Willing to use an acceptable contraceptive method to prevent pregnancy for 3 months after RT.
11. Blood tests values:

    * Leucocytes ≥3000mm3,
    * Absolute neutrophil count ≥1500mm3,
    * Platelets ≥100,000 mm3,
    * Total bilirubin ≤ 1.5xULN,
    * AST, SGOT, SGPT ≤2.5xULN, If Alkaline Phosphatase ≤ 4xULN, then transaminases are normal.
    * Creatinine ≤ 2.0xULN.
    * INR or Prothrombin time ≤1.5xULN.

Exclusion Criteria:

1. Concomitant chemotherapy or immunotherapy within the past 4 weeks
2. Fit for surgical exploration unless the patient refuses surgery
3. Known hypersensitivity to any of the components of the treatment.
4. Patients undergoing systemic immunosuppressive therapy excepting intermittent, brief use of systemic corticosteroids.
5. Longest tumor diameter >7 cm.
6. Clinically significant cardiovascular disease, e.g. cardiac failure of New York Heart Association classes III-IV, uncontrolled coronary artery disease, cardiomyopathy, uncontrolled arrhythmia, uncontrolled hypertension, or history of myocardial infarction in the last 12 months.
7. Patients with uncontrolled intercurrent illnesses including, but not limited to an active infection requiring systemic therapy (not including cholangitis) or a known psychiatric or substance abuse disorder(s) that would interfere with cooperation with the requirements of the trial or interfere with the study endpoints.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Patient requires treatment not specified in this protocol which may conflict with the endpoints of this study including evaluation of response or toxicity of Alpha DaRT.
10. Volunteers participating in another interventional study in the past 30 days which might conflict with the endpoints of this study or the evaluation of response or toxicity of Alpha DaRT.
11. High probability of protocol non-compliance (in opinion of investigator).
12. Breastfeeding women or women of childbearing potential unwilling or unable to use an acceptable contraceptive method to prevent pregnancy for 3 months after RT.
13. Subjects not willing to sign an informed consent

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility - DaRT seed placement | immediately following the insertion procedure
  Feasibility will be determined according to the rate of successful placement of Alpha DaRT
Safety - Adverse events | From day 0
  Safety will be determined according to the overall incidence of device related AEs and SAE's graded according to CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Efficacy -Alpha DaRT seeds | 1, 3, and 6 months post DaRT insertion].
  The study's secondary objective will be to evaluate efficacy, as determined by local control evaluation according to RECIST v1.1

IPD SHARING:
Plan to Share IPD: No